CLINICAL TRIAL: NCT05226052
Title: Effect of the Use of Probiotic Saccharomyces Boulardii on Acute Viral Inflammatory Diarrhea Diagnosed With Multiplex PCR Technique, Randomized Clinical Trial (RCT).
Brief Title: Effect of the Use of Probiotic S. Boulardii on Acute Viral Inflammatory Diarrhea Diagnosed With Multiplex PCR.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, GONZALEZ-OJEDA ALEJANDRO, Clinical Professor, Instituto Mexicano del Seguro Social
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020-PCR-SB
Record Dates: First submitted 2021-12-14; First posted 2022-02-07 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Viral Diarrhea

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: : The person delegated to assigns treatment is the nurse of the medical office. Assignment will be done using a simple excel algorithm. The cans are numbered sequentially. The blindness will be broken until the statistical analysis is completed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- S. boulardii (Experimental): treatment arm group (3 capsules of Floratil 200mg®/day)
  Interventions: Dietary Supplement: Saccharomyces boulardii (Floratil 600mg)
- Placebo (Placebo Comparator): control group (3 capsules of placebo/day)
  Interventions: Dietary Supplement: 3 capsules of placebo

INTERVENTIONS:
Dietary Supplement: Saccharomyces boulardii (Floratil 600mg) — PGIC and PGIS assessment
  Other Names: PGIC and PGIS assessment
  Arms: S. boulardii
Dietary Supplement: 3 capsules of placebo — PGIC and PGIS assessment
  Other Names: PGIC and PGIS assessment
  Arms: Placebo

SUMMARY:
Acute diarrhea (AD) has been a public health problem throughout the history of Mexico. According to the epidemiological surveillance system, between 2008-2017, five to six million new cases of AD occurred per year. Clinical presentation of viral gastroenteritis ranges from an asymptomatic state to diarrhea with severe dehydration. Viral etiology can be difficult to differentiate from those of gastroenteritis caused by enteric bacteria based solely on clinical presentation, especially due to the presence of leukocytes in stool, since it was thought that only diarrhea of bacterial etiology was present and what defines it as acute inflammatory diarrhea; therefore, laboratory studies are essential to make a specific diagnosis. In addition to methylene blue test traditionally performed to describe the presence of leukocytes in stool, multiplex PCR is an automated system in which the extraction, amplification and detection of nucleic acid occurs in a single closed pouch. The panel includes for the etiological identification of bacteria, parasites and viruses. Probiotics are effective for acute infectious diarrhea caused by bacteria, but there are inconsistent results on the effectiveness of probiotics for diarrhea caused by viruses. It is important to note that there are no studies in the adult population with acute diarrhea of viral etiology identified by PCR Multiplex in our environment and the use of probiotics to reduce the period of convalescence. Mexico also lacks for detection tests to identify the pathogen, that can be used routinely in clinical practice, as other countries has shown the economical, clinical outcomes and patient satisfaction results with it. In a review, S. boulardii shows an effectiveness in 4 of the 6 studies where it was used as a treatment in acute adult viral diarrhea, where it was used as a treatment. Based on this review, because it considers the adult population, it will be used S. boulardii as a treatment in patients diagnosed with acute viral diarrhea, to reduce the days of presence of associated symptoms. The Patient Global Impression scale (PGI) is the Patient-reported outcomes counterpart to the Clinical Global Impressions scale. The PGIS are 1-item questionnaire that ask an individual patient to rate the severity of a specific condition at baseline and or to rate at endpoint the perceived change in his/her condition in response to therapy; in the other hand PGIC measures change in clinical status

DETAILED DESCRIPTION:
Acute diarrhea (AD) has been a public health problem throughout the history of Mexico. According to the epidemiological surveillance system, between 2008 and 2017, five to six million new cases of AD occurred per year. The clinical presentation of viral gastroenteritis ranges from an asymptomatic state to diarrhea with severe dehydration. Viral etiology can be difficult to differentiate from those of gastroenteritis caused by enteric bacteria based solely on clinical presentation, especially due to the presence of leukocytes in stool, since it was thought that only diarrhea of bacterial etiology was present and what defines it as acute inflammatory diarrhea; therefore, laboratory studies are essential to make a specific diagnosis. In addition to methylene blue test traditionally performed to describe the presence of leukocytes in stool, Multiplex Polymerase Chain Reaction (PCR) is an automated system in which the extraction, amplification and detection of nucleic acid occurs in a single closed pouch. The panel includes for the etiological identification of bacteria, parasites and viruses. Probiotics are effective for acute infectious diarrhea caused by bacteria, but there are inconsistent results on the effectiveness of probiotics for diarrhea caused by viruses. It is important to note that there are no studies in the adult population with acute diarrhea of viral etiology identified by PCR Multiplex in our environment and the use of probiotics to reduce the period of convalescence. Mexico also lacks for detection tests to identify the pathogen, that can be used routinely in clinical practice, as other countries has shown the economical, clinical outcomes and patient satisfaction results with it. In a review, S. boulardii shows an effectiveness in 4 of the 6 studies where it was used as a treatment in acute adult viral diarrhea, where it was used as a treatment. Based on this review, because it considers the adult population, it wll be used S. boulardii as a treatment in patients diagnosed with acute viral diarrhea, to reduce the days of presence of associated symptoms. The Patient Global Impression scale (PGI) is the Patient-reported outcomes counterpart to the Clinical Global Impressions scale. The Patient Global Impression scale of Severity (PGIS) are 1-item questionnaire that ask an individual patient to rate the severity of a specific condition (single-state scales) at baseline and or to rate at endpoint the perceived change in his/her condition in response to therapy; in the other hand The Patient Global Impression scale of Change (PGIC) measures change in clinical status.

Research question: What is the effect of the use of probiotic S. boulardii on acute inflammatory diarrhea of viral etiology diagnosed with multiplex PCR technique? Hypothesis: The use of S. boulardii in patients with acute viral inflammatory diarrhea diagnosed with the Multiplex PCR technique will decrease the days of associated symptoms and self-reported improvement.

Main objective: To analyze the effect of the use of S. boulardii on acute inflammatory viral diarrhea diagnosed with the Multiplex PCR technique.

Specifics: 1. To determine the incidence of viral pathogens in patients diagnosed with acute inflammatory viral diarrhea treated in the gastroenterology and coloproctology area. 2. To identify the incidence of associated symptoms in both groups in day 4 and 8 after diagnosis. 3. Compare the days of self-reported improvement by the patient between both groups using the PGIS and PGIC surveys.

ELIGIBILITY:
Inclusion Criteria:

* patients who give their informed consent,
* over 18 years of age,
* leukocytes in the stool,
* confirmed diagnosis of viral infection using the multiplex PCR

Exclusion Criteria:

* Confirmed diagnosis of infection by bacteria and/or parasites, associated or not with viral etiology;
* autoimmune diseases or immunosuppressive treatment;
* previous administration of antibiotic treatment during the last 7 days;
* consumption of any type of probiotic in the last 7 days;
* known allergy to probiotic containing S. boulardii;
* Inflammatory Bowel Disease;
* positive test or clinical positivity to the current operational definition for severe acute respiratory syndrome coronavirus 2 (SARS-COV-2).
* patients who do not have medical insurance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2020-12-21 (Actual); Primary Completion 2022-01-03 (Actual); Study Completion 2022-01-03 (Actual)

PRIMARY OUTCOMES:
Number of subjects with S. boulardii on acute inflammatory viral diarrhea diagnosed with Multiplex PCR technique as treatment that have a change in the severity of their symptoms measured with PGIS and PGIC assessments at day 4 and day 8. | 8 days
  The Patient Global Impression scale (PGI) is the Patient-reported outcomes counterpart to the Clinical Global Impressions scale. The PGIS are 1-item questionnaire that ask an individual patient to rate the severity of a specific condition (single-state scales) at baseline and or to rate at endpoint the perceived change in his/her condition in response to therapy; in the other hand PGIC measures change in clinical status.

SECONDARY OUTCOMES:
Number of subjects with acute inflammatory viral diarrhea treated in the gastroenterology and coloproctology area | 365 days
  To determine the incidence of viral pathogens in patients diagnosed with acute inflammatory viral diarrhea treated in the gastroenterology and coloproctology area during the 12 month period; measured by applying the multiplex PCR test to determine the causative pathogen.
Number of subjects presenting associated symptoms in both groups in day 4 and 8 after diagnosis | 8 days
  To identify the incidence of associated symptoms, such as: fever and abdominal pain; assessed using the patient's daily record.

OTHER OUTCOMES:
Compare the days of self-reported improvement by the patient between both groups using the PGIS and PGIC surveys. | 8 days
  Compare the days of self-reported improvement by the patient between both groups using the PGIS and PGIC surveys.

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Gonzalez Ojeda, MD, PhD, Study Director — Instituto Mexica del Seguro Social
Locations (1):
- Hospital Puerta de Hierro Sur, Tlajomulco de Zúñiga, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Savola KL, Baron EJ, Tompkins LS, Passaro DJ. Fecal leukocyte stain has diagnostic value for outpatients but not inpatients. J Clin Microbiol. 2001 Jan;39(1):266-9. doi: 10.1128/JCM.39.1.266-269.2001. PMID 11136781
- [Result] Villarruel G, Rubio DM, Lopez F, Cintioni J, Gurevech R, Romero G, Vandenplas Y. Saccharomyces boulardii in acute childhood diarrhoea: a randomized, placebo-controlled study. Acta Paediatr. 2007 Apr;96(4):538-41. doi: 10.1111/j.1651-2227.2007.00191.x. Epub 2007 Feb 14. PMID 17306006
- [Result] Wang LP, Zhou SX, Wang X, Lu QB, Shi LS, Ren X, Zhang HY, Wang YF, Lin SH, Zhang CH, Geng MJ, Zhang XA, Li J, Zhao SW, Yi ZG, Chen X, Yang ZS, Meng L, Wang XH, Liu YL, Cui AL, Lai SJ, Liu MY, Zhu YL, Xu WB, Chen Y, Wu JG, Yuan ZH, Li MF, Huang LY, Li ZJ, Liu W, Fang LQ, Jing HQ, Hay SI, Gao GF, Yang WZ; Chinese Centers for Disease Control and Prevention (CDC) Etiology of Diarrhea Surveillance Study Team. Etiological, epidemiological, and clinical features of acute diarrhea in China. Nat Commun. 2021 Apr 29;12(1):2464. doi: 10.1038/s41467-021-22551-z. PMID 33927201
- [Result] Pang XL, Preiksaitis JK, Lee BE. Enhanced enteric virus detection in sporadic gastroenteritis using a multi-target real-time PCR panel: a one-year study. J Med Virol. 2014 Sep;86(9):1594-601. doi: 10.1002/jmv.23851. Epub 2013 Nov 14. PMID 24242161
- [Result] Chiejina M, Samant H. Viral Diarrhea. 2023 Sep 5. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK470525/ PMID 29262044
- [Result] Farfan M, Piemonte P, Labra Y, Henriquez J, Candia E, Torres JP. [Filmarray GI TM panel for detection of enteric pathogens in stool samples: preliminary experience]. Rev Chilena Infectol. 2016 Feb;33(1):89-91. doi: 10.4067/S0716-10182016000100016. Spanish. PMID 26965886
- [Result] Olaiz-Fernandez GA, Gomez-Pena EG, Juarez-Flores A, Vicuna-de Anda FJ, Morales-Rios JE, Carrasco OF. [Historical overview of acute infectious diarrhea in Mexico and future preventive strategies]. Salud Publica Mex. 2020 Jan-Feb;62(1):25-35. doi: 10.21149/10002. Spanish. PMID 31869558
- [Result] Palacio-Mejia LS, Rojas-Botero M, Molina-Velez D, Garcia-Morales C, Gonzalez-Gonzalez L, Salgado-Salgado AL, Hernandez-Avila JE, Hernandez-Avila M. Overview of acute diarrheal disease at the dawn of the 21st century: The case of Mexico. Salud Publica Mex. 2020 Jan-Feb;62(1):14-24. doi: 10.21149/9954. PMID 31314211
- [Result] Matthijnssens J, Otto PH, Ciarlet M, Desselberger U, Van Ranst M, Johne R. VP6-sequence-based cutoff values as a criterion for rotavirus species demarcation. Arch Virol. 2012 Jun;157(6):1177-82. doi: 10.1007/s00705-012-1273-3. Epub 2012 Mar 20. PMID 22430951
- [Result] Lanata CF, Fischer-Walker CL, Olascoaga AC, Torres CX, Aryee MJ, Black RE; Child Health Epidemiology Reference Group of the World Health Organization and UNICEF. Global causes of diarrheal disease mortality in children <5 years of age: a systematic review. PLoS One. 2013 Sep 4;8(9):e72788. doi: 10.1371/journal.pone.0072788. eCollection 2013. PMID 24023773
- [Result] Ahmed SM, Hall AJ, Robinson AE, Verhoef L, Premkumar P, Parashar UD, Koopmans M, Lopman BA. Global prevalence of norovirus in cases of gastroenteritis: a systematic review and meta-analysis. Lancet Infect Dis. 2014 Aug;14(8):725-730. doi: 10.1016/S1473-3099(14)70767-4. Epub 2014 Jun 26. PMID 24981041
- [Result] Sniffen JC, McFarland LV, Evans CT, Goldstein EJC. Choosing an appropriate probiotic product for your patient: An evidence-based practical guide. PLoS One. 2018 Dec 26;13(12):e0209205. doi: 10.1371/journal.pone.0209205. eCollection 2018. PMID 30586435
- [Result] Allen SJ, Martinez EG, Gregorio GV, Dans LF. Probiotics for treating acute infectious diarrhoea. Cochrane Database Syst Rev. 2010 Nov 10;2010(11):CD003048. doi: 10.1002/14651858.CD003048.pub3. PMID 21069673
- [Derived] Salazar-Parra MA, Cruz-Neri RU, Trujillo-Trujillo XA, Dominguez-Mora JJ, Cruz-Neri HI, Guzman-Diaz JM, Guzman-Ruvalcaba MJ, Vega-Gastelum JO, Ascencio-Diaz KV, Zarate-Casas MF, Gonzalez-Ponce FY, Barbosa-Camacho FJ, Fuentes-Orozco C, Cervantes-Guevara G, Cervantes-Perez E, Cervantes-Cardona GA, Cortes-Flores AO, Gonzalez-Ojeda A. Effectiveness of Saccharomyces Boulardii CNCM I-745 probiotic in acute inflammatory viral diarrhoea in adults: results from a single-centre randomized trial. BMC Gastroenterol. 2023 Jul 3;23(1):229. doi: 10.1186/s12876-023-02863-8. PMID 37400812